CLINICAL TRIAL: NCT02765529
Title: Research of Biomarkers of Air Pollutants Exposure
Brief Title: Biomarkers of Exposure to Air Pollutants (AEROTOX-2)
Acronym: AEROTOX-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: Universite du Littoral Cote d'Opale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-RT-13; 2015-A00983-46 (Other: ANSM)
Record Dates: First submitted 2016-04-25; First posted 2016-05-06 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Biomarkers of Air Pollution Exposure
Keywords: Environmental Pollution; Fine particles; Biomarkers; Elderly
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 20-30 years (Experimental): Blood sampling
  Interventions: Procedure: Blood sampling
- 45-55 years (Experimental): Blood sampling
  Interventions: Procedure: Blood sampling
- 70-80 years (Experimental): Blood sampling
  Interventions: Procedure: Blood sampling
- Control (Experimental): Blood sampling for standardization of technical procedures
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling

SUMMARY:
Nowadays, an increase of inflammatory chronic diseases and/or tumors incidence has been reported in part due to the rising in life expectancy. For instance, exposure to air pollution, and in particularly to fine particles has been classified by the International Agency for Research on Cancer (IARC) as a risk factor for cancer, being the elderly population particularly sensitive. However, no validated biomarkers have been identified to assess the exposure to fine particles maybe correlated to cancerogenesis.

AEROTOX-2 is a prospective pilot study on the ex vivo effects of the atmospheric pollution exposure. The study aims to identity new biomarkers after an exposure of leukocytes to doses of fine particles.

Secondly, the study aims to analyze, according to age, the leukocytes response to the urban pollution exposure.

DETAILED DESCRIPTION:
To estimate the influence of the atmospheric pollution on the whole adult population, subjects will be recruited in a wide range of age (20 - 80 years).

Samples of atmospheric particles will be collected in Dunkerque (North of France), one of the most important industrial areas in France. This city is influenced by car traffic, urban and industrial activities, and the wide sea traffic of the North Sea. Therefore, Dunkerque is a reference site to study the atmospheric pollution and its impact on health.

These markers will be searched in association with the different mechanisms involved in the toxicity of the fine particles such as: inflammatory response, genotoxicity, metabolic activity and epigenetic changes after exposure of leukocytes isolated from patients to doses of fine particles.

The study of the correlation between biological observations and conditions of exposure to air particles will bring answers about the impact of the environmental pollution on the health of vulnerable populations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-30 years, 45-55 years or 70-80 years
* Signature of an informed consent
* Non-smoker or ex-smoker for more than 10 years
* Homogeneous repartition between men and women
* Social insurance affiliation
* Understanding or being able to speak French

Exclusion Criteria:

* Pregnant or breast feeding woman
* Treatment with parenteral corticoids in the 30 days prior to inclusion visit, treatment with immunosuppressant drugs, radiotherapy, chemotherapy
* Occupational exposure (metallurgy, petrochemistry, house painter) for more than 10 years and having ceased all activities in these areas for less than 10 years ago.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Level of expression of blood biomarkers of air pollution exposure | through the study completion, an average of 48 months
  These markers will be searched in association with the different mechanisms involved in the toxicity of the fine particles such as: inflammatory response, genotoxicity, metabolic activity and epigenetic changes after exposure of leukocytes to doses of fine particles.

SECONDARY OUTCOMES:
Total amount of different populations of peripheral blood leucocytes | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles.
Measure of the expression of genes involved in metabolism by quantitative polymerase chain reaction (qPCR) | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles.
Measure of the expression of genes involved in metabolism by TaqMan Gene Expression Assays | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles.
Detection of genotoxicity by identification of DNA double-strand breaks and DNA adducts | through the study completion, an average of 48 months
Detection of epigenetic modifications | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles. In order to measure the expression of hundreds of miRNAs within a given sample a microarray analysis technology will be performed using the TaqMan® Low Density Array Human MicroRNA.
Correlation between age and markers of inflammation | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles.
Correlation between age and markers of metabolic activity | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles.
Correlation between age and markers genotoxicity | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles.
Correlation between age and markers of epigenetic modifications | through the study completion, an average of 48 months
  After exposure of leukocytes to doses of fine particles.

CONTACTS AND LOCATIONS:
Overall Officials: Gosset Pierre, MD, Principal Investigator — Lille Catholic University; Sylvain Billet, Study Chair — UCEIV
Locations (1):
- Clinical Nutrition Center Naturalpha, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No